CLINICAL TRIAL: NCT05111574
Title: A Randomized Phase II Trial of Adjuvant Nivolumab With or Without Cabozantinib in Patients With Resected Mucosal Melanoma
Brief Title: Using Nivolumab Alone or With Cabozantinib to Prevent Mucosal Melanoma Return After Surgery
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2021-11794; NCI-2021-11794 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); A091903 (Other: Alliance for Clinical Trials in Oncology); A091903 (Other: CTEP); U10CA180821 (NIH)
Record Dates: First submitted 2021-11-05; First posted 2021-11-08 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Anal Melanoma; Bladder Melanoma; Cervical Melanoma; Esophageal Melanoma; Gallbladder Melanoma; Head and Neck Mucosal Melanoma; Mucosal Melanoma; Nasopharyngeal Mucosal Melanoma; Oral Cavity Mucosal Melanoma; Penile Mucosal Melanoma; Rectal Melanoma; Recurrent Mucosal Melanoma; Sinonasal Mucosal Melanoma; Urethral Melanoma; Urinary System Mucosal Melanoma; Vaginal Melanoma; Vulvar Melanoma
MeSH Terms: interventions — Specimen Handling; cabozantinib; Magnetic Resonance Spectroscopy; Nivolumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 (nivolumab, cabozantinib) (Experimental): Patients receive nivolumab IV over 30 minutes on day 1 and cabozantinib PO QD of each cycle. Treatment repeats every 28 days for up to 13 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO during screening and as clinically indicated throughout the trial. Patients may undergo CT, MRI, or PET/CT at baseline, CT and MRI may be repeated every 6 months on study. Additionally, patients may undergo bone scans, as well as optional blood and tissue sample collection throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Drug: Cabozantinib S-malate; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab; Procedure: Positron Emission Tomography
- Arm 2 (nivolumab, placebo) (Active Comparator): Patients receive nivolumab IV over 30 minutes on day 1 and placebo PO QD of each cycle. Treatment repeats every 28 days for up to 13 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO during screening and as clinically indicated throughout the trial. Patients may undergo CT, MRI, or PET/CT at baseline, CT and MRI may be repeated every 6 months on study. Additionally, patients may undergo bone scans, as well as optional blood and tissue sample collection throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab; Drug: Placebo Administration; Procedure: Positron Emission Tomography
- Arm 3 (nivolumab, cabozantinib) (Experimental): Patients receive nivolumab IV over 30 minutes and cabozantinib PO QD of each cycle. Treatment repeats every 28 days for up to 26 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO during screening and as clinically indicated throughout the trial. Patients may undergo CT, MRI, or PET/CT at baseline, CT and MRI may be repeated every 6 months on study. Additionally, patients may undergo bone scans, as well as optional blood and tissue sample collection throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Drug: Cabozantinib S-malate; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood and tissue sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Drug: Cabozantinib S-malate — Given PO
  Other Names: BMS-907351; Cabometyx; Cometriq; XL 184; XL-184; XL184
  Arms: Arm 1 (nivolumab, cabozantinib); Arm 3 (nivolumab, cabozantinib)
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
Drug: Placebo Administration — Given PO
  Arms: Arm 2 (nivolumab, placebo)
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT

SUMMARY:
This phase II trial tests whether nivolumab in combination with cabozantinib works in patients with mucosal melanoma. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Cabozantinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It works by blocking the action of an abnormal protein that signals tumor cells to multiply. This helps stop the spread of tumor cells. Giving nivolumab in combination with cabozantinib could prevent cancer from returning.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the efficacy of adjuvant nivolumab (480 mg every [q]4 weeks) versus nivolumab plus cabozantinib s-malate (cabozantinib) (40 mg daily) in patients with mucosal melanoma.

SECONDARY OBJECTIVES:

I. To compare overall survival between the two adjuvant therapies. II. To evaluate the adverse effects in each arm. III. To assess the correlation between PD-L1 expression in tumor cells with survival (recurrence free survival [RFS] and overall survival [OS]).

IV. To evaluate the overall response rate (ORR), duration of response (DOR), progression free survival (PFS), and OS of nivolumab plus cabozantinib in patients who cannot undergo gross total resection of disease or have metastatic disease at baseline.

V. Results of the primary analysis will be examined for consistency, while taking into account the stratification factors and/or covariates of baseline quality of life (QOL) and fatigue.

OUTLINE: Patients whose tumor has been fully removed by surgery are randomized to Arm 1 or Arm 2. Patients whose tumor has not been fully removed by surgery or has spread are assigned to Arm 3.

ARM 1: Patients receive nivolumab intravenously (IV) over 30 minutes on day 1 and cabozantinib orally (PO) once daily (QD) of each cycle. Treatment repeats every 28 days for up to 13 cycles in the absence of disease progression or unacceptable toxicity.

ARM 2: Patients receive nivolumab IV over 30 minutes on day 1 and placebo PO QD of each cycle. Treatment repeats every 28 days for up to 13 cycles in the absence of disease progression or unacceptable toxicity.

ARM 3: Patients receive nivolumab IV over 30 minutes and cabozantinib PO QD of each cycle. Treatment repeats every 28 days for up to 26 cycles in the absence of disease progression or unacceptable toxicity.

Patients undergo echocardiogram (ECHO) during screening and as clinically indicated throughout the trial. Patients may undergo computed tomography (CT), magnetic resonance imaging (MRI), or positron emission tomography (PET)/CT at baseline, CT and MRI may be repeated every 6 months on study. Additionally, patients may undergo bone scans, as well as optional blood and tissue sample collection throughout the trial.

After completion of study treatment, patients are followed up every 3 months until disease progression, and then every 6 months for up to 5 years from registration or until death.

ELIGIBILITY:
Inclusion Criteria:

* STEP 0 INCLUSION CRITERIA
* Histologically proven mucosal melanoma by local pathology
* Central PD-L1 tumor tissue submission
* STEP 1 INCLUSION CRITERIA
* Receipt of the central PD-L1 testing results available

  * Report is required for randomization of resection R0 or R1 patients
  * Testing must be started in Step 0 but results can be reported after registration for resection R2 patients
* Disease status-Resected R0 or R1 disease patients. Patients eligible for randomization have resected R0 or R1 disease (with negative margins or positive microscopic margins) that must meet one of the following 4 criteria as defined below:

  * Regional lymph node (LN) involvement; OR
  * In-transit metastases/satellite primary disease; OR
  * Single localized, primary disease meeting one of the following site-specific requirements:

    * Head/neck - Sinonasal (including nasopharynx): any primary lesion; Nasal or oral cavity; pT4a or above, given slightly improved OS

      * NOTE: Conjunctival: does not meet the qualification for eligibility
    * Anorectal - any primary lesion
    * Vaginal/cervical - any primary, as they have 5 year OS rates of 5-25%
    * Urinary tract - any primary urethral or bladder tumor
    * Penile
    * Vulvar- American Joint Committee on Cancer (AJCC) cutaneous stage IIB or higher
    * Esophageal/gallbladder - any primary
  * Locoregionally recurrent following prior resection, meeting at least one of the above criteria
  * In addition, patients must have undergone cross-sectional imaging of the brain, chest, abdomen and pelvis with no evidence of distant metastatic disease
* Disease status-Non-resected R2 or metastatic disease patients

  * Non-resected R2 or metastatic disease that is assessable and measurable radiographically or by physical examination
* Prior Treatment:

  * No prior systemic checkpoint inhibitor therapy of mucosal melanoma, including in the adjuvant setting, is allowed. Prior adjuvant chemotherapy or interferon is allowed.
  * No other active, concurrent malignancy that requires ongoing systemic treatment or interferes with radiographic assessment of melanoma response as determined by the investigator. Exceptions may allow for adjuvant no evidence of disease (NED) cancers undergoing hormone based therapy may be eligible pending the other eligibility criteria are met and the principal investigator (PI) affirms the hormonal agent would not change the melanoma response.
  * Any radiation must have completed 28 days prior to randomization and the patient must have adequately recovered from its effects.
  * For resectable patients only: Surgery must have completed 28 days prior to randomization.
  * For resectable patients only: Surgery must have completed no more than 84 days prior to randomization.
* Not pregnant and not nursing, because this study has an agent that has known genotoxic, mutagenic and teratogenic effects. Therefore, for women of childbearing potential only, a negative pregnancy test done =< 7 days prior to registration is required
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Creatinine =< 1.5 x upper limit of normal (ULN) OR creatinine clearance (CrCl) >= 50mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Albumin >= 2.8 g/dL
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 x upper limit of normal (ULN)
* No cardiovascular disease, including:

  * No history of acute coronary syndromes (including myocardial infarction and unstable angina), coronary artery bypass graft (CABG) coronary angioplasty, or stenting within 6 months prior to study entry.
  * No history of current class II or higher congestive heart failure as defined by the New York Heart Association (NYHA) functional classification system.
  * No refractory hypertension defined as a blood pressure of systolic > 140 mmHg and/or diastolic > 90 mmHg despite adequate attempts at anti-hypertensive therapy.
  * No history of myocarditis.
  * No history of syncope of cardiovascular etiology, uncontrolled cardiac arrhythmia, history of Mobitz II second degree or third degree heart block without a permanent pacemaker in Association (NYHA) class II to IV heart failure, or stroke/transient ischemic attack (TIA) within the past 3 months.
  * No corrected QT interval by Fridericia's formula (QTcF) > 500 msec. Note: if initial QTcF is found to be > 500 ms, two additional electrocardiograms (EKGs) separated by at least 3 minutes should be performed. If the average of these three consecutive results for QTcF is =< 500 ms, the subject meets eligibility in this regard.
* No underlying hematologic issues, including:

  * Congenital bleeding diathesis
  * Gastrointestinal (GI) bleeding requiring intervention within the past 6 months, unless directly related to mucosal melanoma
  * Active hemoptysis within 42 days prior to study enrollment.
  * Active tumor lesions with cavitations or tumor lesions which invade, encase, or abut major blood vessels. The anatomic location and characteristics of primary tumors or metastases as well as the medical history should be carefully reviewed in the selection of subjects for treatment with cabozantinib/placebo.
  * Pulmonary emboli or deep vein thromboses (DVT) that require an active anticoagulation regimen.
  * No known or suspected history of cytopenia (low white blood cell [WBC], hemoglobin or platelet count) of greater than 3 months duration with an unknown cause, myelodysplastic syndrome, or hematologic malignancies.
* No clinical, laboratory or radiographic evidence of an active bacterial, fungal, or viral infection requiring treatment at the time of pre-registration (e.g., active symptoms of COVID-19 infection or a post-infectious symptomatic autoimmune syndrome, serious bacterial infections requiring antibiotics).
* No known or suspected gastrointestinal disorder affecting absorption of oral medications.
* Comorbid conditions:

  * No active autoimmune disease or any condition requiring systemic treatment with either corticosteroids (> 10 mg daily of prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
  * No history of autoimmune motor neuropathy (e.g., Guillain-Barre syndrome, myasthenia gravis) or non-infectious pneumonitis.
  * No history of severe allergic reactions to an unknown allergen or any components of the study drugs or its excipients.
  * No history of gastrointestinal perforation or abdominal fistula.
  * No clinically suspected central nervous system (CNS) (leptomeningeal or parenchymal) metastases. Patients with a history of CNS metastasis(s) will be allowed as long as

    * The metastatic site(s) were adequately treated as demonstrated by clinical and radiographic improvement, AND
    * The patient has recovered from the intervention (no residual adverse events > Common Terminology Criteria for Adverse Events [CTCAE] grade 1), AND
    * The patient has remained without occurrence of new or worsening CNS symptoms for a period of 28 days prior to enrollment.
  * No history of seizure or any condition that may increase the patient's seizure risk (e.g., prior cortical stroke, significant brain trauma) within 2 years.
  * No clinically active or chronic liver disease resulting in moderate/severe hepatic impairment (Child-Pugh class B or C), ascites, coagulopathy or bleeding due to liver dysfunction.
  * No untreated spinal cord compression or evidence of spinal metastases with a risk of impending fracture or spinal cord compression. Spinal metastases must have completed planned radiation or surgical therapy prior to registration.
* Concomitant medications:

  * Chronic concomitant treatment with strong inhibitors of CYP3A4 is not allowed on this study. Patients on strong CYP3A4 inhibitors must discontinue the drug for 5 days prior to the start of study treatment.
  * Chronic concomitant treatment with strong CYP3A4 inducers is not allowed. Patients must discontinue the drug 5 days prior to the start of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2022-08-11 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence free survival (RFS) | Number of days from registration until either local or distant recurrence or death (due to any cause), assessed up to 5 years
  Will evaluate RFS of single agent adjuvant nivolumab plus placebo compared to the combination treatment of adjuvant nivolumab plus cabozantinib in patients with resected mucosal melanoma.

SECONDARY OUTCOMES:
Overall survival (OS) | Number of days from registration until death (due to any cause, assessed up to 5 years
  Will be evaluated utilizing the Kaplan-Meier (KM) method and, when appropriate, cox proportional hazards models. Median OS is calculated (along with 95% Confidence intervals) using the KM method. A Cox proportional hazards model is built to compare arms 1 and 2 with respect to OS.
RFS | Number of days from registration until either local or distant recurrence or death (due to any cause), assessed up to 5 years
  Median RFS will be calculated (along with 95% Confidence intervals) using the KM method. A Cox proportional hazards model will also be built to compare arms 1 and 2 with respect to RFS, with and without stratifying for PD-L1 categorization. For non-resected cohort, If a patient in this group has surgery, their RFS data will be censored at the time of surgery.
Progression free survival | Number of days from registration until either radiographic or clinical progression or death (due to any cause), assessed up to 5 years
  Will be evaluated in multiple settings utilizing the KM method and, when appropriate, cox proportional hazards models.
Objective response rate (Arm 3) | Up to 5 years
  Will assess this endpoint utilizing a two-stage Simon that looks to improve from a rate of 20% to 47%.
Duration of response (Arm 3) | Time from the first evidence of response until progression, assessed up to 5 years
  A KM analysis is performed to calculate the median duration of response and 95% confidence intervals are constructed.
Incidence of adverse events | Up to 5 years
  The maximum grade for each type of adverse event will be summarized using Common Terminology Criteria for Adverse Events version 5.0. The frequency and percentage of grade 3+ adverse events will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander N Shoushtari, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (147):
- United States (143):
  - Sutter Auburn Faith Hospital, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Keck Medicine of USC Koreatown, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Mills Health Center, San Mateo, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - The Melanoma and Skin Cancer Institute, Englewood, Colorado
  - UM Sylvester Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Bronson Battle Creek, Battle Creek, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo Cancer Center, Kalamazoo, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Hematology Oncology Associates of CNY at Camillus, Camillus, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Miami Valley Hospital South, Centerville, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - M D Anderson Cancer Center, Houston, Texas
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sheboygan, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
- Canada (4):
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm